CLINICAL TRIAL: NCT02867462
Title: Information Consultation by a Manipulator Radiotherapy: Impact on Information to Patients Treated With Radiotherapy for Cancer
Brief Title: Information Consultation by Radiotherapy Manipulator
Acronym: INFORTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012/63 INFORTH; 2012-A01601-42 (Other: ANSM ID RCB)
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2016-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-Standard Care (Other): standard care
  Interventions: Other: Standard care
- B-manipulator consultation radiotherapy added to standard care (Experimental): manipulator consultation radiotherapy added to standard care
  Interventions: Other: manipulator consultation radiotherapy added to standard care

INTERVENTIONS:
Other: Standard care — standard care
  Arms: A-Standard Care
Other: manipulator consultation radiotherapy added to standard care
  Arms: B-manipulator consultation radiotherapy added to standard care

SUMMARY:
The medical teams are increasingly sought by patients to get the most possible information, probably expressed in a different form and thereby supplementing the information already received. Coulter et al. reached similar conclusions in their study of the writings of patient information documents. They point out, moreover, the best adaptation of the patients better informed compared to those with less or no information.

This need for information varies over time. It is present before treatment begins, continues during treatment and persists after treatment. Given the specific features of radiotherapy, the manipulators are important interlocutors to participate in the accompanying caregiver time.

In conclusion, the quality of information delivered to the patient has been poorly evaluated, let alone with validated tools in this area.

The impact of information on the tolerance of the treatment also needs to be confirmed, knowing that an informed patient seems less anxious and better prepared for future treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer of the head and neck, esophagus, stomach, breast, rectum, anal canal, prostate, lung, bile duct, pancreas or female genital histologically proven
* Patient being treated by radiotherapy alone or combined with chemotherapy / immunotherapy, exclusive treatment or adjuvant
* Age over 18 years

Exclusion Criteria:

* Patient has been treated with radiation to the tumor site
* Patient with metastatic stage disease
* Patient targeted for hypofractionated radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ-INFO25 | 12 weeks
  amount of information received by patients in the case of a standard support and if the patient has a consultation with a radiation therapy manipulator, assessed using the questionnaire EORTC QLQ-INFO25 before the first radiotherapy session

CONTACTS AND LOCATIONS:
Overall Officials: Karen BENEZERY, md, Principal Investigator — Centre Antoine Lacassagne
Locations (1):
- Centre Antoine LACASSAGNE, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided